CLINICAL TRIAL: NCT04473846
Title: The Use of Propofol-fentanyl-ketamine (PFK) Combination Versus General Anesthesia Using Propofol and Fentanyl in Patients Undergoing Endoscopic Procedures: a Prospective Study
Brief Title: Propofol-fentanyl-ketamine (PFK) Combination Versus General Anesthesia Using Propofol and Fentanyl in Patients Undergoing Endoscopic Procedures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Abdelkarim Saleh AlOweidi, Principal Investigator, University of Jordan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 67/2020/524
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Anesthesia
Keywords: Anesthesia; Endoscopy; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PF group (Experimental): The first group will undergo general anesthesia using Fentanyl and Propofol.
  Interventions: Drug: PK general anesthesia
- PFK group (Experimental): The second group will receive a mixture that consists of Fentanyl, Propofol, and Ketamine. In addition, Lidocaine will be added to reduce the pain on injection caused by Propofol.
  Interventions: Drug: PFK combination

INTERVENTIONS:
Drug: PK general anesthesia — Patients will be anesthetized using Fentanyl (2 mcg/kg) and Propofol (1-2 mg/kg).
  Arms: PF group
Drug: PFK combination — Each patient received an initial dose of 0.05 ml/kg from the solution, then after waiting for 60 seconds, another 0.05 ml/kg were given. Maintenance was given as boluses of 0.025 ml/kg every three to five minutes.
  Arms: PFK group

SUMMARY:
Conscious sedation provides adequate control of pain and anxiety for the majority of routine endoscopic procedures as well as adequate amnesia. Sedation practices vary widely, with some colonoscopists advocating sedation only for the most difficult cases of colonoscopy, while others prefer using deep sedation or general anaesthesia for colonoscopy. However, many physicians are still using moderate sedation for the majority of patients.

The use of propofol, a short acting anesthetic agent, for conscious sedation provides a considerably more rapid onset of action and shorter recovery time, for which it is believed to be a safe drug of choice for patients undergoing endoscopic procedures. Although propofol cannot be used as a single agent for moderate sedation, it can be effectively titrated to moderate sedation after administration of small doses of narcotics and sedatives.

The aim of this study is to compare between general anesthesia and deep sedation using propofol-fentanyl-ketamine (PFK) preparation in terms of perioperative vital signs, intraoperative awareness, post-operative pain scores, and the use of analgesia postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients who were admitted for endoscopic and colonoscopic procedures.
* ASA (American Society of Anaesthesiologists physical status) score from 1 to 3.

Exclusion Criteria:

* patient refusal.
* urgent and emergency cases, which were not elective procedures.
* Surgeries that were expected to take a long duration (more than 1.5 hour).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Transient decrease in oxygen saturation | 1 hour
  the investigators will record any episodes of transient reduction of oxygen saturation.
Blood pressure stability | 1 hour
  the investigators will record changes in blood pressure after induction of anesthesia
Recovery time | 2 hours
  the investigators will document recovery time in the post anesthesia care unit (PACU) until recovery of full consciousness.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan